CLINICAL TRIAL: NCT02076243
Title: Phase II Trial of Nab-Paclitaxel as First Line Cytotoxic Chemotherapy in Patients With Unresectable and Metastatic Cutaneous Squamous Cell Carcinoma
Brief Title: Treatment With Nab-paclitaxel in Cutaneous SCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed by sponsor
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Philip Friedlander, Assistant Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1697
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: cutaneous squamous cell carcinoma; SCC; abraxane; nab-paclitaxel; unresectable; metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nab-paclitaxel (Experimental): weekly dosed nab-paclitaxel chemotherapy (days 1, 8 , 15 of a 28 day cycle) administered as an I.V. infusion over approximately 30 minutes. Dosage is determined by weight and height of participant.
  Interventions: Drug: nab-paclitaxel

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel (abraxane) administered weekly (days 1,8, and 15 of 28 day cycle) to patients with unresectable locoregional or distantly metastatic cutaneous squamous cell carcinoma (SCC).
  Other Names: abraxane

SUMMARY:
This is an investigator initiated phase II study to assess the efficacy of a chemotherapy called nab-paclitaxel as first line cytotoxic chemotherapy in subjects with unresectable locally advanced or metastatic cutaneous squamous cell carcinoma (SCC). All subjects receive the treatment by vein weekly and receive the same dose of the treatment.

The risk of developing cutaneous SCC is approximately 10% in a lifetime. The vast majority are treated surgically and do not recur. However a small percentage become unresectable over time or metastasize distantly in the body. Unresectable and metastatic cutaneous SCC has a poor prognosis and oncologists often choose a whole body therapy without the benefit of prospective efficacy data. Very little prospective investigation into the efficacy of specific chemotherapy regimens as a function of line of therapy has been performed in this patient population. Nab-paclitaxel is type of chemotherapy that has demonstrated activity in other types of cancer such as lung and head and neck cancers. The primary objective of this study is to determine the response rate (percentage of subjects with tumor shrinkage) to nab-paclitaxel treatment in subjects with cutaneous SCC who have not received cytotoxic chemotherapy in the unresectable or the metastatic settings.. Secondary objectives are the progression free survival (time until tumor starts to grow), safety, assessment of the percentage of subjects whose tumor expresses a protein called SPARC, and correlating the expression of SPARC with response to treatment. To determine if the tumor expresses SPARC part of a prior standard biopsy such as that performed to establish the diagnosis of SCC will be used. SPARC is a protein that is overexpressed in a range of different cancer types and may alter the environment around the tumor possibly in a way that may make the SCC more responsive to treatment with nab-paclitaxel.

DETAILED DESCRIPTION:
Non-melanoma skin cancers represent the most common type of cancer in the United States with cutaneous SCC comprising 20% of these malignancies. The risk of developing cutaneous SCC is approximately 10% in a lifetime. This risk increases with age and varies according to the latitude in which one lives. The incidence rate in the United States is increasing as a result of multiple factors including altered sun exposure patterns and population aging. Early detection is critical as the vast majority are cured by definitive localized therapy with an overall 5-year cure rate of greater than 90%.

Although the vast majority of cutaneous SCCs are treated surgically with curative intent the estimated case fatality rate ranges from 1-5% depending on reported study. If regional lymph nodes are involved a standard treatment approach is lymphadenectomy followed by the consideration of adjuvant therapy (radiation +/- chemotherapy). However a subset of these patients ultimately will develop unresectable or distantly metastatic recurrences.

Unresectable SCC is treated using systemic approaches usually encompassing cytotoxic chemotherapy. However clinical investigation to determine efficacy of specific agents has been very limited and not studied in a rigorous fashion. Efficacy data stems largely from case reports and limited case series and from a very small number of phase II trials. As for targeted therapies, treatment with cetuximab demonstrated limited activity (RR 11%) in a 36 patient phase II trial. Many oncologists tend to treat with platinum agents, taxanes and 5-FU based regimens. However no standard exists. As such there is a need to explore more systematically the efficacy of specific chemotherapeutic agents with the goal of developing a standard treatment approach.

Nab-paclitaxel is an intriguing option to use for treatment given demonstrated efficacy in other malignancies with SCC histology. In clinical practice many oncologists use paclitaxel despite the lack of rigorous clinical investigation. The use of paclitaxel is limited by toxicities associated with the solvent Cermaphor EL.

Nab-paclitaxel is an albumin bound form of paclitaxel. In other malignancies such as breast cancer nab-paclitaxel is associated with improved response rates and time to progression relative to paclitaxel. Nab-paclitaxel based chemotherapy has demonstrated efficacy in other malignancies with SCC histology including head and neck carcinoma and NSCLC.

SPARC (secreted protein acidic and rich in cysteine), also known as osteonectin and BM-40, is a 43kD secreted extracellular matrix glycoprotein first identified in 1984 and noted to have high binding affinity for albumin. SPARC further affects angiogenesis by interacting with growth factors such as VEGF and basic fibroblast growth factor (bFGF). It binds with platelet derived growth factor (PDGF) inhibiting binding to its receptors. SPARC interacts with bFGF and inhibits the migration of endothelial cells.

Overexpression of SPARC has been found in many tumor types including breast, melanoma, brain, colon, skin and several others and is associated with increased tumor invasion and metastasis. For example, in melanoma SPARC expression is clinically correlated with aggressiveness and metastatic phenotypes. In melanoma models SPARC is associated with decreased E-cadherin and increased N-cadherin expression, suggesting that it may regulate epithelial-mesenchymal transition in the earlier stages of malignant transformation. SPARC expression has also been associated with increased breast cancer cell invasiveness. The absence of SPARC has been shown to suppress the development of UV-induced squamous cell carcinoma in a mouse model.

Another tumor promoting mechanism of SPARC is in its interaction with inflammation. There is evidence that SPARC may play a role in dampening the immune response to tumor cells. Melanoma cells lacking SPARC expression induced neutrophil recruitment, increased chemotactic factors such as IL-8, GRO, and leukotrienes and resulted in tumor cell rejection. This observation decreased neutrophil recruitment in the presence of SPARC has also been noted in other models including SPARC null versus wild type mice. SPARC may regulate the apoptotic pathway of neutrophils involving Fas ligand.

SPARC is able to affect tumor progression at several levels. It plays a role in epithelial-mesenchymal transformation. It promotes tumor growth and metastasis by inhibiting immune surveillance and promoting angiogenesis and it is correlated with metastatic cell aggressiveness.

The overexpression of SPARC in many tumors and the tumor microenvironment and its high binding affinity for albumin make an albumin-bound drug delivery attractive. Via the gp60 and caveolae-mediated albumin transport pathway albumin is transported from the blood vessel into the tumor. Albumin-bound paclitaxel (nab-paclitaxel) was approved by the FDA in January 2005 for the treatment of metastatic breast cancer. Nab-paclitaxel takes advantage of this transport carrying paclitaxel into tumor cells. There it may be preferentially retained in tissues overexpressing SPARC. SPARC has been shown to be overexpressed in squamous cell carcinomas of the head and neck (61%, versus 0% in normal head and neck tissue).

The use of intra-arterial nab-paclitaxel has been examined in locally advanced squamous cell carcinoma of the head and neck with response rates of 75-78%. A retrospective analysis showed that SPARC upregulation in the tumor tissue was associated with increased response in 16 patients with squamous cell carcinoma of the head and neck who received intra-arterial nab-paclitaxel.

This is a single arm phase II study assessing the efficacy of treatment with nab-paclitaxel (abraxane) administered weekly (days 1,8, and 15 of 28 day cycle) to patients with unresectable locoregional or distantly metastatic cutaneous squamous cell carcinoma (SCC). A Simon 2 stage design will be used. If no responses are seen in the first 12 patients it will be concluded that the response rate is no greater than 3% and the trial will be stopped for futility at the end of stage one. Otherwise the trial will enroll 9 more patients for a total of 21.

In summary, the development of unresectable locally advanced or distantly metastatic cutaneous SCC confers a very poor prognosis. While various types of systemic therapy are used by oncologists choices are based on anecdotal experiences and a limited number of case series and small phase II studies. Nab-paclitaxel has demonstrated significant anti-tumor activity in several malignancies of SCC morphology. Taxanes are often used as systemic treatment for unresectable cutaneous SCC. This study will allow for prospective evaluation of the activity of abraxane as first line systemic cytotoxic chemotherapy (a defined line of cytotoxic therapy) in the treatment of advanced SCC. The hypothesis of this phase II study is that abraxane will demonstrate significant anti-tumor activity a defined by a primary endpoint of best overall response rate. It is hypothesized that increased SPARC expression will correlate with response to nab-paclitaxel treatment and serve as a biomarker for treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable locoregional or distantly metastatic squamous cell carcinoma arising from a cutaneous surface, lip, or ear. Basosquamous histology is eligible.
* ECOG PS 0 or 1
* Life expectancy of more than 4 months
* Adequate renal, hepatic, and bone marrow function:
* Patients must have adequate liver function: AST and ALT < 2.5 X upper limit of normal, alkaline phosphatase < 2.5 X upper limit of normal, unless bone metastasis is present in the absence of liver metastasis, Bilirubin < 1.5 mg/dL
* Patients must have adequate bone marrow function: Platelets >100,000 cells/mm3, Hemoglobin > 9.0g/dL, WBC > 3,000 cells/mm3, and ANC > 1,500 cells/mm3
* Patients must have adequate renal function: creatinine <1.5 mg/dL
* Age > 18 years old
* Women of childbearing potential and sexually active males must agree to use effective contraception during treatment and for three months after completing treatment
* Negative serum or urine B-hCG pregnancy test at screening for patients of childbearing potential
* No previous or concurrent malignancy except inactive nonmelanoma skin cancer, in situ carcinoma of the cervix, treated grade 1 papillary bladder cancer, localized prostate cancer detected via biopsy only and being treated with "watchful waiting", or other cancers where the patient has no evidence of recurrence for more than 5 years
* Must be at least 28 days since surgical procedure and/or radiation therapy and at least 4 weeks since last treatment with targeted therapies such as cetuximab or immunotherapy.
* No significant inter-current illness such as serious infection requiring intravenous antibiotics.
* Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE v4.0)
* Ability to provide informed consent

Exclusion Criteria:

* Prior systemic cytotoxic chemotherapy for unresectable SCC. Prior adjuvant or neoadjuvant cytotoxic chemotherapy provided not within prior 28 days is allowed. Prior systemic therapies with a targeted agent (cetuximab) or immunotherapy in the setting of unresectable SCC (is allowed).
* Prior taxane based chemotherapy
* The presence of any CNS tumor that has not been stable for at least 3 months off of corticosteroids and confirmed by imaging.
* Prior major organ transplant or autoimmune disease requiring chronic immunosuppression
* Psychiatric illness or social situation that would preclude compliance.
* Active or chronic infection with HIV, hepatitis B or hepatitis C. Formal testing should be performed if clinical suspicion.
* Patients with New York Heart Association class II, III, or IV disease or arrhythmia requiring treatment (rate controlled Atrial fibrillation is allowed)
* Lack of measurable disease on imaging studies as defined by RECIST 1.
* Any condition that in the opinion of the treating physician is likely to prevent the patient from complying with any aspect of the protocol or that may put the patient at unacceptable risk
* Known allergy to treatment medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Friedlander, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nab-paclitaxel
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: the percentage of subjects who develop Complete Response (CR) or Partial Response (PR)
Time Frame: at week 8 post treatment
Population: study terminated, results not collected
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 0

2. Secondary Outcome: Median Progression Free Survival
Description: every eight weeks will reassess efficacy by imaging and can continue treatment if no progression and expect will be up to an average 5 years
Time Frame: average 5 years
Population: study terminated, results not collected
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Prevalence of SPARC Expression
Description: prevalence of SPARC expression in advanced squamous cell cancer of the skin. The tumor specimen used to determine SPARC expression wll be obtained from a biopsy previously performed as standard of care (such as to establish the diagnosis).
Time Frame: at baseline
Population: study terminated, results not collected
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 0

4. Secondary Outcome: Treatment Response
Description: correlation of response to first line treatment with Nab-Paclitaxel with SPARC expression, with target lesions measured at the longest diameter of each non-lymph node lesion and the short axis for target lymph nodes
Time Frame: at week 8 post treatment
Population: study terminated, results not collected
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety and Tolerability
Description: number of participants with adverse events as a measure of safety and tolerability
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Arm/Group | Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel (N=2)
Sepsis (Infections and infestations) | 1 (1)
Fall (General disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel (N=2)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbumenia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain Right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes